CLINICAL TRIAL: NCT06237907
Title: The Role of Pyroptosis and Ferroptosis in the Pathophysiology of Lymphedema
Brief Title: Pyroptosis and Ferroptosis in the Pathophysiology of Lymphedema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201327B0
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-09

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent surgery
  Interventions: Other: Patients underwent lymphedema surgery; Other: Patients underwent surgery without LVA

INTERVENTIONS:
Other: Patients underwent lymphedema surgery — Patients who have developed lymphedema and undergone lymphedema surgery.
Other: Patients underwent surgery without LVA — For patients who have not experienced lymphedema but require surgery due to other disease such as cancer, trauma, chronic wounds, skin defects, etc.

SUMMARY:
The project aims to compare the differences in the expression of cell death through apoptosis and iron-dependent cell death after the reduction of edema symptoms following lymphedema surgery in patients.

DETAILED DESCRIPTION:
This project aims to investigate the expression of cell death through apoptosis and iron-dependent cell death in the subcutaneous adipose tissue of patients with lymphedema. The study also seeks to explore the roles of these processes among lymphatic endothelial cells, adipocytes, and macrophages, and their association with lymphedema, thus gaining insights into the pathophysiological mechanisms of lymphedema. Furthermore, the project aims to compare the differences in the expression of cell death through apoptosis and iron-dependent cell death after the reduction of edema symptoms following lymphedema surgery in patients.

ELIGIBILITY:
Inclusion Criteria:

* Control Group: Patients who have not experienced lymphedema but require surgery due to other diseases such as cancer, trauma, chronic wounds, skin defects, etc.
* Experimental Group: Patients who have lymphedema and undergone lymphedema surgery.

Exclusion Criteria:

* 1. Individuals with venous thrombosis, chronic heart failure, and renal failure.
* 2. Vulnerable populations, individuals with limited mobility, pregnant women, and minors.
* 3. Those expected to be unable to attend follow-up visits or complete the study smoothly.
* 4. Participants who express doubts about the trial and cannot provide satisfactory answers.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients as experimental group who has lymphedema and need to underwent surgery. Patients as control group who require surgery without lymphedema. Written informed consent was obtained from all patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
The correlation between post-LVA volume reduction | 1 month after surgery
  The differences in expression of cell necrosis and iron-dependent cell death after lymphedema surgery were observed in patients, following alleviation of edema symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan